CLINICAL TRIAL: NCT05632315
Title: A Phase II Randomized Trial to Evaluate the Impact of Fecal Microbiota Transplantation Using the Penn Microbiome Therapy Products on Recipient and Environmental Colonization With Multidrug-Resistant Organisms
Brief Title: PMT for MDRO Decolonization
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 852552
Record Dates: First submitted 2022-11-17; First posted 2022-11-30 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Multidrug Resistant Bacterial Infection; Enterobacteriaceae Infections; Pseudomonas Aeruginosa; VRE Infection; Methicillin-resistant Staphylococcus Aureus
MeSH Terms: conditions — Enterobacteriaceae Infections; Pseudomonas Infections

STUDY DESIGN:
Intervention Model Description: Randomized, open label, comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (24):
- ESCRE/CRE BL-BLI (Experimental): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: Beta Lactamase Inhibitors (BL-BLI)
  Interventions: Drug: PMT
- ESCRE/CRE BL-BLI standard of care (SOC) (No Intervention): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: Beta Lactamase Inhibitors (BL-BLI) standard of care (SOC)
- ESCRE/CRE carbapenem +/- BLI (Experimental): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: carbapenem +/- BLI
  Interventions: Drug: PMT
- ESCRE/CRE carbapenem +/- BLI standard of care (SOC) (No Intervention): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: carbapenem +/- BLI standard of care (SOC)
- ESCRE/CRE Fluoroquinolone (Experimental): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: Fluoroquinolone
  Interventions: Drug: PMT
- ESCRE/CRE Fluoroquinolone standard of care (SOC) (No Intervention): MDRO: extended-spectrum cephalosporin resistant Enterobacterales ESCRE/CRE Antibiotic Class: Fluoroquinolone standard of care (SOC)
- MRSA lipo/glycopeptide (Experimental): MRDO: methicillin-resistant S. aureus (MRSA) Antibiotic Class: lipo/glycopeptide
  Interventions: Drug: PMT
- MRSA lipo/glycopeptide standard of care (SOC) (No Intervention): MRDO: methicillin-resistant S. aureus (MRSA) Antibiotic Class: lipo/glycopeptide standard of care (SOC)
- MRSA oxazolidinone (Experimental): MRDO: methicillin-resistant S. aureus (MRSA) Antibiotic Class: oxazolidinone
  Interventions: Drug: PMT
- MRSA oxazolidinone standard of care (SOC) (No Intervention): MRDO: methicillin-resistant S. aureus (MRSA) Antibiotic Class: oxazolidinone standard of care (SOC)
- MDR-PA BL-BLI (Experimental): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: Beta Lactamase Inhibitors (BL-BLI)
  Interventions: Drug: PMT
- MDR-PA BL-BLI standard of care (SOC) (No Intervention): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: Beta Lactamase Inhibitors (BL-BLI) standard of care (SOC)
- MDR-PA carbapenem +/- BLI (Experimental): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: carbapenem +/- BLI
  Interventions: Drug: PMT
- MDR-PA carbapenem +/- BLI standard of care (SOC) (No Intervention): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: carbapenem +/- BLI standard of care (SOC)
- MDR-PA Fluoroquinolone (Experimental): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: Fluoroquinolone
  Interventions: Drug: PMT
- MDR-PA Fluoroquinolone standard of care (SOC) (No Intervention): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: Fluoroquinolone standard of care (SOC)
- VRE lipopeptide (Experimental): MDRO: vancomycin resistant Enterococcus (VRE) Antibiotic Class: lipopeptide
  Interventions: Drug: PMT
- VRE lipopeptide standard of care (SOC) (No Intervention): MDRO: vancomycin resistant Enterococcus (VRE) Antibiotic Class: lipopeptide standard of care (SOC)
- VRE oxazolidinone (Experimental): MDRO: vancomycin resistant Enterococcus (VRE) Antibiotic Class: oxazolidinone
  Interventions: Drug: PMT
- VRE oxazolidinone standard of care (SOC) (No Intervention): MDRO: vancomycin resistant Enterococcus (VRE) Antibiotic Class: oxazolidinone standard of care (SOC)
- ESCRE/CRE cefepime/cefidericol (Experimental): MDRO: ESCRE/CRE Antibiotic Class: cefepime/cefidericol
  Interventions: Drug: PMT
- ESCRE/CRE cefepime/cefidericol standard of care (SOC) (No Intervention): MDRO: ESCRE/CRE Antibiotic Class: cefepime/cefidericol standard of care (SOC)
- MDR-PA cefepime/cefidericol (Experimental): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: cefepime/cefidericol
  Interventions: Drug: PMT
- MDR-PA cefepime/cefidericol standard of care (SOC) (No Intervention): MDRO: two-class non-susceptible Pseudomonas aeruginosa (MDR-PA) Antibiotic Class: cefepime/cefidericol standard of care (SOC)

INTERVENTIONS:
Drug: PMT — Fecal Microbiota for Transplant, enema product (PMT-001) or Fecal Microbiota for Transplant, suspension product (PMT-002)
  Other Names: Penn Microbiome Therapy
  Arms: ESCRE/CRE BL-BLI; ESCRE/CRE Fluoroquinolone; ESCRE/CRE carbapenem +/- BLI; ESCRE/CRE cefepime/cefidericol; MDR-PA BL-BLI; MDR-PA Fluoroquinolone; MDR-PA carbapenem +/- BLI; MDR-PA cefepime/cefidericol; MRSA lipo/glycopeptide; MRSA oxazolidinone; VRE lipopeptide; VRE oxazolidinone

SUMMARY:
This is a randomized, open label, comparative Phase II trial being conducted to determine whether fecal microbiota transplant using Penn Microbiome Therapy (PMT) products helps standard therapy eradicate antibiotic-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Multidrug-resistant organism (MDRO) infection of the bloodstream, respiratory tract, or urinary tract. Qualifying MDROs include extended-spectrum cephalosporin-resistant Enterobacterales (ESCRE) or carbapenem-resistant Enterobacterales (CRE), Pseudomonas aeruginosa non-susceptible to two or more classes of antibiotics (MDR-PA), vancomycin-resistant Enterococcus (VRE), and methicillin-resistant Staphylococcus aureus (MRSA).
2. On appropriate antibiotic treatment per clinical phenotypic susceptibility testing of the qualifying MDRO, and with a qualifying antibiotic class. Qualifying antibiotic classes include beta-lactam + beta-lactamase inhibitor, carbapenem (with or without betalactamase inhibitor), fluoroquinolone, lipopeptide, glycopeptide, or oxazolidinone.
3. Expected duration of inpatient antibiotic treatment for index MDRO infection at least 5 days total.
4. At least two calendar days remaining, and no more than 7 calendar days remaining prior to SCAIM (scheduled completion of inpatient appropriate antibiotics for the index MDRO infection).
5. Age ≥ 18 years.

Exclusion Criteria:

1. Evidence of colon/small bowel perforation at the time of study screening.
2. Unable to tolerate enteral and enema nutrition and medication administration (i.e., only able to tolerate intravenous nutrition and medications).
3. Goals of care are directed to comfort rather than curative measures.
4. Moderate or severe neutropenia within 10 calendar days prior to enrollment.
5. Known food allergy that could lead to anaphylaxis.
6. Known allergy to fecal microbiota transplant products or their components
7. Pregnancy or lactation

   1. For subjects of childbearing potential (ages 18 to 55) and who are randomized to receive the intervention, the subject must have a negative pregnancy test within 24 hours prior to product administration
   2. Female or male subjects (ages 18 to 55) of reproductive potential engaged in active sexual activity that could lead to a pregnancy must agree to use one of the following forms of birth control while receiving study medications and through day 28 following completion of treatment, at minimum:

   i. Male or female condoms

   ii. Diaphragm or cervical cap with spermicide, if available

   iii. Intrauterine device (IUD)

   iv. Oral contraceptives or other hormonal contraception
8. Known gastrointestinal disease that could affect the safety of fecal microbiota transplant at time of enrollment:

   1. Inflammatory Bowel Disease (IBD)
   2. Short Gut Syndrome
   3. Fistulas
   4. Bowel resection surgery
   5. Colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with resolution of index MDRO colonization of the gut | 30 (+/-7)- day visit after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
  measured by selective stool culture, resolution will be defined as the absence of growth of the index MDRO on selective culture media.
Frequency of solicited adverse events (AEs) | randomization until 180 day visit after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Frequency of serious adverse events (SAEs) | randomization until 180 day visit after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Frequency of adverse events of special interest (AESIs) | randomization until 180 day visit after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Frequency of medically attended adverse events (MAAEs) | randomization until 180 day visit after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)

SECONDARY OUTCOMES:
Eradication of gut colonization with the index MDRO | 7 days and 90 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
  i.e., negative selective bacterial culture for the index MDRO to be assessed in addition to primary endpoint
Eradication of gut colonization with any of the included MDROs | 7- , 30-, and 90-days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
All-cause mortality | 30- and 60-days following SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Colectomy occurrence | within 30 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Cumulative days of hospitalization | from randomization to 30 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Cumulative days of intensive care | from randomization to 30 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Bacteria growth in blood samples | from randomization to 30 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Hospital admission | within 60 days of discharge from index hospitalization
Hospital admission | within 180 days after SCAIM (scheduled completion of appropriate inpatient antibiotics for the index MDRO infection)
Instances of worsened abdominal pain, fever, tachycardia, and hypotension | randomization until 180-day visit
Instances of aspiration (including reduced oxygen saturation, tachypnea, or respiratory distress (PMT-002 upper entral delivery only) | randomization until 180-day visit
Instances of fever, diarrhea, nausea and vomiting | 7-, 30-, 90- and 180 day follow up visits
Instances of new metabolic disease, including hyperglycemia, thyroid disease, weight gain or loss | 30-, 90- and 180 day follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Brendan J Kelly, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Emory University - Grady Memorial Hospital, Atlanta, Georgia
  - Washington University, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No